CLINICAL TRIAL: NCT07211906
Title: Effects of Oral Nursing Education on Oral Health and Quality of Life in Patients With Home Non-Invasive Ventilator
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202500853B0
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-07

CONDITIONS: Oral Health Care; Oral Hygiene; Noninvasive Ventilators; Sleep Quality; Quality of Life
Keywords: Oral health; Oral hygiene; Noninvasive ventilation; Quality of Life; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants receive routine oral care guidance or standard education materials without additional digital support or structured intervention. This group serves as a baseline to evaluate the effectiveness of the tailored oral health education and digital follow-up.
  Interventions: Other: Control Group: oral hygiene education standard
- Intervention (Experimental): The intervention group in this study received a structured oral care program integrated with technological support via Line communication. Specifically, participants in the experimental group were provided with personalized oral hygiene guidance through one-on-one oral care instruction, which included oral health education and demonstration. They also received continuous support and follow-up through the Line communication platform, where they could reply to educational prompts and clarify doubts, fostering adherence to oral care practices over a three-month period. This approach aimed to improve oral health outcomes and quality of life among home non-invasive ventilation users through a combination of direct guidance and digital communication.
  Interventions: Other: Control Group: oral hygiene education standard; Other: oral hygiene education program

INTERVENTIONS:
Other: Control Group: oral hygiene education standard — oral hygiene education Standard care: oral hygiene education standard care, which involved providing participants with printed oral health education leaflets without additional personalized instruction or digital support. Specifically, participants were assessed at baseline, and then, at one-month intervals, they received printed oral care instructions and completed follow-up assessments. This group was not provided oral education or interactive guidance via digital platforms during the study period.
Other: oral hygiene education program — Oral hygiene education program:
  The oral hygiene education program includes a "Line-based oral care guidance program," which involves personalized, one-on-one oral health education facilitated through the Line communication platform. The process began with an initial pre-test assessment, including interviews and questionnaire evaluations. Then, the participants engaged in the "Line-guided oral care" intervention, where they received tailored guidance and demonstrated
  Arms: Intervention

SUMMARY:
This study evaluated the impact of oral care guidance on oral health and quality of life in patients using non-invasive ventilation at home. Using a randomized controlled trial, results showed significant improvements in oral hygiene, overall health, sleep quality, and daily living after the intervention. Additionally, better oral care was positively associated with enhanced sleep quality and overall well-being. The findings suggest that targeted oral health education can effectively improve the health and quality of life for home non-invasive ventilation users, supporting its integration into clinical practice.

DETAILED DESCRIPTION:
This study focused on exploring how providing specific oral care guidance can benefit individuals who rely on non-invasive ventilation (NIV) at home. Non-invasive ventilation is a respiratory support method used by people suffering from chronic respiratory conditions, such as COPD (chronic obstructive pulmonary disease), to help them breathe more easily without the need for invasive procedures like intubation.

The research aimed to see whether improving oral hygiene through targeted education could positively impact these patients' oral health, sleep quality, and overall quality of life. Since poor oral health has been linked to respiratory infections and other health complications, the study hypothesized that better oral care might help reduce related problems and enhance daily living.

In the study, participants receiving NIV at home were divided into two groups: one received comprehensive oral health guidance and education tailored to their needs, while the control group continued with usual care without additional instruction. The intervention included instructions on proper oral hygiene practices, such as effective brushing and oral cleaning, tailored to the specific needs of NIV users, and was provided over a period of three months.

Throughout the study, the researchers collected data on various aspects including oral health status, sleep quality, and overall life satisfaction. They used validated questionnaires like the Pittsburgh Sleep Quality Index (PSQI) to evaluate sleep and the Oral Health Impact Profile-14 (OHIP-14) to assess oral health-related quality of life.

The results demonstrated that patients who received the oral care guidance showed significant improvements in their oral health, sleep quality, and overall well-being compared to those in the control group. The intervention not only helped with maintaining better oral hygiene but also contributed to a better sleep experience and higher quality of life, reducing the negative impacts associated with respiratory diseases and the challenges of long-term NIV use.

Importantly, implementing such educational programs in clinical settings can empower patients to take better care of their oral health, which in turn may reduce the risk of infections and other complications, ultimately improving their daily lives. The study highlights the importance of integrating oral health education into the routine care for patients with chronic respiratory conditions on home NIV, emphasizing a holistic approach to patient health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants aged 18 years or older with full legal capacity. 2. Able to communicate in Mandarin or Taiwanese. 3. Currently using a non-invasive ventilator. 4. Individuals with natural dentition or complete edentulism will be included. 5. Able to operate and use the LINE communication application.

Exclusion Criteria:

- 1. Individuals who are unable to independently comprehend or respond to questions.

2. Individuals whose daily living activities rely on caregiver assistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Oral Health Assessment Tool (OHAT) | The time frame for measuring outcomes in this study spans four assessment points: baseline (M0), and follow-up at one month (M1), two months (M2), and three months (M3) after the intervention.
  his measure evaluates various aspects of oral health, such as lips, tongue, gingiva, saliva, natural teeth, dentures, oral cleanliness, and pain, with higher scores indicating poorer oral health. The study aims to determine if the oral health education intervention can significantly improve or maintain oral health status over the three-month period

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | The time frame for measuring outcomes in this study spans four assessment points: baseline (M0), and follow-up at one month (M1), two months (M2), and three months (M3) after the intervention.
  This measure evaluates various aspects of sleep over the past month, including sleep quality, latency, duration, efficiency, disturbances, medication use, and daytime dysfunction. Higher PSQI scores indicate poorer sleep quality over the three-month period.

OTHER OUTCOMES:
Chinese version of the SF-12 health survey | The time frame for measuring outcomes in this study spans four assessment points: baseline (M0), and follow-up at one month (M1), two months (M2), and three months (M3) after the intervention.
  daily functioning, providing a comprehensive evaluation of the intervention's effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University Of Science and Technology, Chiayi City, Taiwan, Taiwan